CLINICAL TRIAL: NCT06283303
Title: A Clinical Study to Evaluate the Safety and Efficacy of Herpes Virus T3011 Injection in Combination With Toripalimab and Regorafenib in Patients With Liver Metastases From Colorectal Cancer
Brief Title: A Clinical Study of T3011 in Combination With Toripalimab and Regorafenib in Patients With Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: Immvira Co., Limited (Unknown)
Responsible Party: Principal Investigator, Funan Liu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-HAI-01
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: oncolytic virus; colorectal Cancer; liver metastasis; hepatic artery infusion
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab; regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy with T3011 hepatic artery infusion , Regorafenib and Toripalimab (Experimental): The study was divided into two dose groups, T3011 3×10^8 plaque forming unit(PFU)/time (HAI) and T3011 1×10^9 PFU/time (HAI), with a 3+3 dose escalation design. After the completion of the lead-in period, the patient entered the combination therapy period（combination therapy with T3011 hepatic artery infusion , Regorafenib and Toripalimab）,and the dosage of T3011 was determined according to the safety observation results of the lead-in period, the dose of toripalimab was 80mg intravenously, and regorafenib was 80mg orally once a day.
  Interventions: Biological: T3011 hepatic artery infusion; Drug: toripalimab; Drug: regorafenib

INTERVENTIONS:
Biological: T3011 hepatic artery infusion — The study was divided into two dose groups, T3011 3×10^8 PFU/time (HAI) and T3011 1×10^9 PFU/time (HAI), with a 3+3 dose escalation design. After the completion of the lead-in period, the patient entered the combination therapy period（combination therapy with T3011 hepatic artery infusion , Regorafenib and Toripalimab）,and the dosage of T3011 was determined according to the safety observation results of the lead-in period, the dose of toripalimab was 80mg intravenously, and regorafenib was 80mg orally once a day.
Drug: toripalimab — The combination therapy period: toripalimab, 80mg intravenous ,D2 and D16, 4 weeks per cycle
Drug: regorafenib — The combination therapy period: regorafenib ,80mg orally once a day, D1-D21,4 weeks per cycle

SUMMARY:
This is a phase I, open-label clinical study of T3011 in combination with Toraplizumab and Regorafenib in patients with liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
This trial is a prospective, open-label, investigator-initiated clinical study in patients with liver metastasis from colorectal cancer, aiming to evaluate the safety and efficacy of T3011 herpes virus injection alone or in combination with toripalimab and regorafenib in patients with liver metastasis from colorectal cancer. In this study, the lead-in period of T3011 and the combination therapy period were designed, and the 3+3 dose escalation design was carried out in the lead-in period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥18 years at the time of signing the Informed Consent Form (ICF);
2. Patients with a definitive histopathological or cytological diagnosis of colorectal cancer with hepatic metastases who have received and failed at least second-line standard therapy in the past, or who have been assessed by the investigator to be unsuitable for standard therapy;
3. Patients with at least one measurable lesion (as defined by RECIST v1.1) that has not been previously treated with radiotherapy (unless definite progression of the lesion has occurred after radiotherapy);
4. Eastern Cooperative Oncology Group(ECOG) score 0 or 1;
5. Expected survival ≥ 12 weeks;
6. For female subjects with childbearing potential, a negative serum pregnancy test within 7 days prior to the first dose of study drug; Acceptance of using medically accepted and effective contraception for at least 6 months after signing the ICF and until the last dose of study drug;
7. Male subjects with childbearing potential agree to use medically accepted and effective contraception from the date of signing the ICF to the date of at least 6 months after the last dose; in addition, the male subject must agree that he will not donate sperm during this period;
8. Understand and voluntarily sign a written ICF and be willing to comply with all trial requirements.

Exclusion Criteria:

1. Patients allergic to the study drug (including its components) or other similar products;
2. Patients who have been treated with oncolytic virus therapy, interleukin-12 (IL-12) in combination with anti PD-1/ PD-L1;
3. Patients who have not recovered from the adverse reactions of previous treatments (the treatment-related toxicity ≤ grade 2, except for alopecia, fatigue or other tolerable events judged by the investigator);
4. Patients with brain metastases that have progressed within 3 months prior to study drug administration (brain metastases that have stabilised within 3 months may be included);
5. History of other malignancies (except cured basal cell skin cancer, cervical carcinoma in situ, papillary thyroid cancer, etc.) within 5 years prior to study drug administration;
6. Patients who received any antineoplastic drug (including but not limited to chemotherapy, biologics, herbal preparations, etc.) within 4 weeks or 5 half-lives (whichever is shorter) prior to study drug administration;
7. Severe hepatic dysfunction (Child Pugh class C), or significant jaundice, hepatic encephalopathy, refractory pleural effusion, or hepatorenal syndrome; Coagulation: international normalized ratio (INR) or Prothrombin time (PT) > 1.5 x Upper limits of normal(ULN) ; activated partial thromboplastin time (aPTT)> 1.5 x ULN; Current comorbidity with active hepatitis: persistent or active hepatitis B (i.e. HBsAg positive or hepatitis B virus (HBV) DNA ≥ upper limit of detection), hepatitis C (HCV RNA ≥ upper limit of detection)] or other hepatitis; Haematology: white blood cell count (WBC) < 3.0 x 10^9/L; platelets < 75 x 10^9/L; haemoglobin < 80g/L; Renal function: serum creatinine >1.5 ULN or creatinine clearance <60 mL/min (Cockcroft-Gault formula calculation)
8. Serious or uncontrollable cardiac disease requiring treatment, congestive heart failure classified as grade 3 or 4 by the New York Heart Association (NYHA), unstable angina not controlled by medication, history of myocardial infarction within 6 months prior to enrolment, serious arrhythmia requiring medication (except atrial fibrillation or paroxysmal supraventricular tachycardia); History of arterial thromboembolic event, venous thromboembolic event of grade ≥3 as defined in NCI CTCAE 5.0, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to randomisation; Current major vascular disease such as aortic aneurysm, aortic coarctation aneurysm, etc. that may be life-threatening or require surgery within 6 months;
9. Previous immunotherapy (including but not limited to PD-1/PD-L1) with immune-related pneumonitis or ≥ grade 3 other immune-related adverse reactions; Current active immune disease requiring systemic treatment with immunosuppressive agents (excluding autoimmune diseases such as vitiligo that do not require intervention, or hypothyroidism that only needs hormone replacement therapy), or immune disease requiring systemic treatment with immunosuppressive agents (e.g., systemic lupus erythematosus) that is likely to recur; Patients with other diseases currently requiring systemic immunosuppressive therapy;
10. HIV Positive; Patients who are currently in the midst of an episode of orofacial herpes; Clinically significant infection or infection treated with intravenous antibiotics within 4 weeks prior to dosing;
11. Inability to swallow, malabsorption syndrome, or uncontrollable nausea, vomiting, diarrhoea or other gastrointestinal disorders that would seriously interfere with drug administration and absorption;
12. Patients who need anti-herpes simplex virus medications (including, but not limited to, acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir, etc.) for the duration of the study, with the exception of topical applications;
13. History of seizures within 12 months prior to study drug administration;
14. Patients with the history of drug use or a history of substance abuse (including alcohol) within one year prior to signing the ICF;
15. Pregnant or lactating women;
16. Other reasons judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event（TEAE） | Complete records until 30 days after the end-of-trial visit (i.e. end of treatment or early termination visit)
  An adverse event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Imaging was performed after completion of the introductory period, i.e. at week 4, and tumour assessment was performed every 8 weeks during the subsequent combined treatment period，assessed up to 100 months
  Objective response rate (ORR) as assessed by the investigators
Overall survival (OS) | Every 3 months until consent withdraw, death, withdrawal study, or loss of follow-up, assessed up to 100 months
  The time from the start of treatment to death for any cause
Progression-free survival (PFS) | Every 8 weeks until disease progression, consent withdraw, death or end of study, assessed up to 100 months
  The time from the start of treatment to progress diease or death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy